CLINICAL TRIAL: NCT01343017
Title: Increased Tidal Volume During Anaesthesia Compared to PEEP. Impact on Arterial Concentration of Sevoflurane, Oxygenation and Cardiac Output in a Randomised Clinical Study of Overweight Patients.
Brief Title: Impact of Increased Tidal Volumes on Oxygenation and Cardiac Output
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Bengt Roth, M.D. , Ph.D., Head of Department, Department of Intensive and Perioperative Care, Lund University Hospital, SE-221 85 Lund, Sweden
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: Dnr 2009/533; EPN 2009/533 (Registry Identifier: Regional Ethics Committee, Lund, Sweden)
Record Dates: First submitted 2011-04-26; First posted 2011-04-27 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-04

CONDITIONS: Obesity
Keywords: Anaesthesia; Pulmonary gas exchange; Functional residual capacity; Cardiac output; Sevoflurane
MeSH Terms: conditions — Obesity | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Increased tidal volume (IVT) (Other): In the group with increased tidal volume (IVT), initial plateau pressure (Pplateau) will be monitored and then tidal volume will be increased until Pplateau was 0.04 cm H2O/kg over the initial Pplateau. The PETCO2 will be then adjusted to 4.5 kPa with a flexible corrugated hose placed between the Y-piece of the anaesthesia circle system and the heat and moisture filter (HME) attached to the endotracheal tube.
  Interventions: Other: Ventilatory pattern
- Normal tidal volume (NVT), with PEEP (Other): In the group with normal tidal volume (NVT), a PEEP to10 cmH2O will be applied. When required, VT will then adjusted to maintain PETCO2 at 4.5 kPa
  Interventions: Other: Ventilatory pattern

INTERVENTIONS:
Other: Ventilatory pattern — In group one, increased tidal volume with a adjusted apparatus dead space volume (IVT), In group two, normal tidal volume with a PEEP to 10 cmH2O applied(NVT). PETCO2 will be adjusted to maintain at 4.5 kPa, in both groups. When PETCO2 values were stable at 4.5 kPa, sevoflurane administration will be started with a vaporiser set to 3%. After 5 minutes the fresh gas flow will be adjusted to 1.0 L/min with an unchanged vaporiser setting throughout the anaesthesia period.
  Other Names: Increased tidal volume (IVT); Normal tidal volume with PEEP (NVT)

SUMMARY:
General anaesthesia impairs respiratory function in overweight patients. The investigators wanted to compare arterial concentration of sevoflurane and oxygen in overweight patients ventilated with increased tidal volume, or normal tidal volume with added 10 cm H2O PEEP.

DETAILED DESCRIPTION:
Functional residual capacity (FRC) and pulmonary gas exchange decrease during induction of general anaesthesia due to closure of airways and genesis of atelectasis. It has been demonstrated that there is a correlation between body constitution and airway closure under general anaesthesia with mechanical ventilation. In the supine position, FRC and respiratory compliance decrease more with an increased body mass index (BMI). In morbidly obese patients general anaesthesia and paralysis lead to even more atelectasis and an increased risk of hypoxemia. In about 90 % of all patients ventilated without positive end-expiratory pressure (PEEP) atelectases are formed, which contribute to impairment of gas exchange. Atelectasis formation can be reduced by PEEP but increasing intrathoracic pressure with PEEP, impairs the venous return to the heart, which reduces stroke volume and cardiac output.

In previous studies the investigators compared the effects of increased tidal volume (VT) with zero end-expiratory pressures (ZEEP) on oxygenation and arterial concentrations of sevoflurane. The investigators found moderately improved oxygenation and a reduced difference between arterial and exhaled carbon dioxide tension with larger tidal volumes achieved this way. The results were similar to what could be expected from an increase in FRC and also included a more efficient uptake of sevoflurane. The investigators have recently confirmed these findings also in overweight patients.

In the present study the investigators will compare arterial concentration of sevoflurane and oxygen in patients with BMI over 25 kg/m2 undergoing abdominal surgery, ventilated with larger tidal volumes or added 10 cmH2O PEEP. The investigators also will assess the influence of these ventilation modes on cardiac output.

Method Ethical approval for this study according to the standards set in the Helsinki declaration (Regional Ethics Committee Dnr: 2009/529 and additions to the application with the measurement of cardiac output Dnr 2010/481) will be provided by Regional Ethics Committee, Lund, Sweden on September 2009 and September 2010. The investigation will include 60 patients, ASA physical status 1 or 2, scheduled for elective colon surgery. Patients will be considered for inclusion in the trial if they will be over 18 yr age and have a BMI more than 25 kg/m2. All procedures will be estimated to last more than 60 minutes. Consent to participate in the study will be received from each patient. Patients with known pulmonary or cardiovascular disease will be excluded. Patients will be randomised to one of two groups with 30 patients in each group via randomly mixed sealed envelope assignment at the start of the procedure in the operating theatre. Interim analysis will be performed after 15 + 15 patients.

Experimental procedure Before start of anaesthesia, an unused carbon dioxide absorber will be applied (Drägersorb, Dräger Medical, Lübeck, Germany) to the anaesthesia ventilator (Dräger Primus™, Dräger Medical, Lübeck, Germany). All patients will be preoxygenated with 100% oxygen for 3-4 minutes with a fresh gas flow of 5 liters/minute. Anaesthesia will be induced with 2 µg/kg fentanyl and 1.5-3.0 mg/kg propofol. Rocuronium 0.6 mg/kg will be administered for muscle paralysis. Ventilation will be assisted manually with 100% oxygen via a semiopen circle system (4.5 L volume) until tracheal intubation and then by means of a ventilator with an FiO2 at 0.35 in nitrogen. The respiratory rate will be 15/min throughout the study and VT will be adjusted as to achieve a PETCO2 at 4.5 kPa. No positive end-expiratory pressure (PEEP) will be applied. Propofol 8 mg/kg/h will be infused until an arterial cannula have been inserted in the radial artery. Stroke volume (SV) and cardiac output (CO) will be assessed in 20 patients (10 in each group) with LIDCO Rapid® (LiDCO Ltd, Cambridge, UK). Transoesophageal echocardiography (TEE) will be used to assess cardiac output in 6 patients (3 in each group) with Philips CX-50®, TEE ultrasound X7-2t (Philips Ultrasound, Bothell, WA, USA). After a control (time zero) sample of arterial blood (3 ml) have been obtained, the ventilatory mode will be altered as follows: In the group with increased tidal volume (IVT), initial plateau pressure (Pplateau) will be monitored and then VT will be increased until Pplateau will be 0.04 cm H2O/kg over the initial Pplateau. The PETCO2 will be then adjusted to 4.5 kPa with a flexible corrugated hose (disposable plastic tube, Medcore, AB Uppsala, Sweden) placed between the Y-piece of the anaesthesia circle system and the heat and moisture filter (HME) attached to the endotracheal tube. This flexible corrugated hose increased the dead-space volume and provided adjustable rebreathing of carbon dioxide. In the group with normal tidal volume (NVT), a PEEP to10 cmH2O will be applied. When required, VT will be then adjusted to maintain PETCO2at 4.5 kPa. In both groups, inspiratory:expiratory ratio was 1:2 including an inspiratory plateau of 10%. When PETCO2 values will be stable at 4.5 kPa, sevoflurane administration will be started with a vaporiser (sevoflurane Dräger Vapor 2000: Medical, Lübeck, Germany) set to 3%. After 5 minutes the fresh gas flow will be adjusted to 1.0 L/min with an unchanged vaporiser setting throughout the anaesthesia period.

Blood samples of 3 ml were drawn from the arterial line into heparinised syringes at 1, 3, 5, 10, 15, 30, 45 and 60 minutes after the start of the sevoflurane administration (totally 27 ml). Arterial oxygen tension (PaO2), oxygen saturation (SaO2) and carbon dioxide tension (PaCO2) will be analysed using an automatic blood gas analyzer (ABL 725™, Radiometer, Copenhagen Denmark). Sevoflurane concentration will be analysed with gas chromatography (GC) on a Perkin-Elmer 3920 gas liquid chromatograph, as previously described.

Patients will be monitored with three-lead ECG, heart rate, oxygen saturation, as measured by pulse oximeter (SpO2) and invasive arterial blood pressure (Solar 8000, General Electric Medical System, Milwaukee, WI, USA). SV and CO were assessed with a LIDCO Rapid® via the arterial catheter. Inspiratory and expiratory oxygen partial pressure (FiO2, PETO2), sevoflurane inspiratory and expiratory partial pressure (Fisevo, PETsevo) and carbon dioxide inspiratory and expiratory partial pressure (FiCO2, PETCO2) will be analysed by the ventilator. Total ventilation per minute, tidal volumes and airway pressures as peak pressure, plateau pressure and mean pressure were measured and documented at the same intervals. Static compliance of the respiratory system will be calculated as tidal volume divided by the inspiratory plateau pressure minus PEEP.

Extra doses of fentanyl (50-100 µg) will be given if mean arterial blood pressure (MAP) increased more than 20% above the initial baseline level. Hypotension (MAP less than 60 mmHg) will be treated with 5-10 mg norepinephrine intravenously. All patients received 3-5 ml/kg/h of glucose solution 2.5% with sodium (70 mmol/l), chloride (45 mmol/l) and acetate (25 mmol/l) intravenously. Neuromuscular blockade will be monitored with a neuromuscular transmission analyzer (TOF-Watch™; Organon Technology B V., Boxel Netherlands). Additional doses of rocuronium were given at the discretion of the anaesthetist.

LiDCO The LiDCO System is a cardiac output monitoring apparatus that uses pulse waveform contour analysis via an arterial catheter. The device uses a proprietary algorithm to analyze the pulse contour by using patient specific data from the patient monitor.16 Linton and colleagues found a good conformity between thermodilutions and LiDCO measurements in 40 patients, with a linear regression value of 0.94.

Transoesophageal echocardiography Stroke volume, cardiac output, and right ventricular function will be assessed using transoesophageal echocardiography. Four and 5-chamber transgastric views will be obtained in all six patients included for TEE. The velocity time integral at the left ventricular outflow tract (VTI LVOT) was measured using pulsed wave Doppler. The diameter of the aorta will be measured using a mid-oesophageal long axis view at the level of the aortic annulus. Measurement of stroke volume will be made by multiplying the LVOT VTI and the aortic diameter. Cardiac output will be calculated by multiplying stroke volume with heart rate. All images will be recorded in triplicate by the same operator and measurements made off-line in a blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1 or 2
* Scheduled for elective colon surgery
* Body mass index more than 25 kg/m2

Exclusion Criteria:

* Patients with known pulmonary or cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Increased tidal volumes impact on sevoflurane and oxygenation | 60 - 90 minutes

SECONDARY OUTCOMES:
Increased tidal volumes impact on cardiac output | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Bodelsson, Professor, Study Chair — Department of Anaesthesia and Intensive Care, Faculty of Medicine, Lund University, Sweden
Locations (1):
- Department of Anaesthesia and Intensiv Care, Faculty of Medicine Lund University, Lund, Lund, Sweden

REFERENCES:
- [Background] Enekvist B, Bodelsson M, Sturesson LW, Johansson A. Larger tidal volume increases sevoflurane uptake in blood: a randomized clinical study. Acta Anaesthesiol Scand. 2010 Oct;54(9):1111-6. doi: 10.1111/j.1399-6576.2010.02291.x. PMID 20887413
- [Background] Enekvist BJ, Luttropp HH, Johansson A. The effect of increased apparatus dead space and tidal volumes on carbon dioxide elimination and oxygen saturations in a low-flow anesthesia system. J Clin Anesth. 2008 May;20(3):170-4. doi: 10.1016/j.jclinane.2007.09.013. PMID 18502358
- [Background] Luttropp HH, Johansson A. Soda lime temperatures during low-flow sevoflurane anaesthesia and differences in dead-space. Acta Anaesthesiol Scand. 2002 May;46(5):500-5. doi: 10.1034/j.1399-6576.2002.460505.x. PMID 12027842
- [Background] Sturesson LW, Johansson A, Bodelsson M, Malmkvist G. Wash-in kinetics for sevoflurane using a disposable delivery system (AnaConDa) in cardiac surgery patients. Br J Anaesth. 2009 Apr;102(4):470-6. doi: 10.1093/bja/aep019. Epub 2009 Feb 25. PMID 19244261